CLINICAL TRIAL: NCT06134245
Title: HOme USability Evaluation
Acronym: HOUSE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS ID: 336920
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Entia Liberty — Home monitoring

SUMMARY:
To validate the usability and safety of the Liberty Analyser.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing systemic anti-cancer therapy (SACT)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, 2 at enrolment
* Adequate English language skills (not requiring a translator) to participate in participant training and use the Entia Liberty analyser
* Patients capable of providing written informed consent

Exclusion Criteria:

* History or current diagnosis of haematological malignancy
* Patients with eyesight or hearing limitations or other disabilities that preclude the use of the Entia Liberty analyser or participation in training
* Inadequate use and understanding of the English language, requiring a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of solid tumour cancer, who are currently undergoing systemic anti-cancer therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The Entia Liberty Analyser is easy to use | Through study completion, 1 day
  Users can easily carry out a test using the Entia Liberty Analyser
The Entia Liberty Analyser is safe to use | Through study completion, 1 day
  Results obtained using the Entia Liberty Analyser are valid and reliable

IPD SHARING:
Plan to Share IPD: Undecided